CLINICAL TRIAL: NCT04449627
Title: Psychological Impact of Admission With Covid-19 During the SARS-CoV-2 Pandemic: Naturalistic Cohort Study With a Digital Intervention
Acronym: FeelGood
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: RoyalFreeNHS
Record Dates: First submitted 2020-06-11; First posted 2020-06-29 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Anxiety Disorders; Post Traumatic Stress Disorder; Depressive Disorder; Covid19
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depressive Disorder; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Naturalistic cohort: Patients who were hospitalised between March and June from Covid19, who did not require treatment in intensive care, who at 8 weeks post discharge have symptoms of anxiety or depression. All patients are offered access to an audio based self help programme based on applied relaxation and mindfulness based cognitive therapy.
  Interventions: Other: Feeling Good Digital App

INTERVENTIONS:
Other: Feeling Good Digital App — Audio based tracks using Jacobson relaxation and mindfullness based cognitive therapy (MBCT) techniques including positive visualisation.

SUMMARY:
Studies have shown that admission to hospital during a coronavirus epidemic is associated with increased levels of anxiety, depression and panic disorder. During the SARS-CoV-2 pandemic in North London the Royal Free Hospital admitted over 500 patients with Covid-19. As part of the standard of care, these patients are screened at 8 weeks post discharge for signs of anxiety and depression. The Feeling Good app is a NHS approved digital application which utilises applied relaxation, mindfulness based cognitive therapy and positive visualisation through audio tracks for the treatment of anxiety and depression.

This is a naturalistic cohort study aimed to track the post illness psychological symptoms of those who have been admitted with Covid-19 to the Royal Free hospital up to 5-7 months after discharge. The study population is those who are exhibiting anxiety or depressive symptoms as measure by the PHQ-2 or TSQ questionnaires. All those with symptoms will be offered free access to a NHS approved app for anxiety and depression, and followed up for 3 months after recruitment to track changes to their symptoms.

DETAILED DESCRIPTION:
It is important that the long-term wellbeing of patients who have been admitted with Covid-19 during the pandemic is addressed. A newly published meta analysis (Rogers et al 2020) has looked at the neuropsychiatric consequences of all coronavirus epidemics, including Serious Acute Respiratory Syndrome (SARS) and Middle East Respiratory (MERS) outbreaks, as well as the first emerging studies from SARS-CoV-2. These studies demonstrate that postillness neuropsychiatric complications including anxiety and depression can persist up to 36 months after the original illness. This is a naturalistic cohort trial with a digital intervention. The study population consists of those patients who were admitted with Covid-19, during the SARS-CoV-2 pandemic, who at 8 weeks after discharge were found to have symptoms relating to anxiety and depression. In this context Covid-19 refers to the disease caused by the virus (named SARS-CoV-2). The study population does not include those who required intensive care admission during their stay. Excluding usual community psychiatric services (for example improving access to psychological therapies) and some specialist intensive care follow up services, no interventions at the Royal Free have been set up to address the long-term psychological impacts of admission to hospital with COVID-19. The digital intervention is an app that consists of twelve audio tracks that combine applied relaxation, mindfulness, cognitive behaviour therapy and positive visualisation. It is a validated guided self-help tool for treatment of anxiety and depression in the NHS, and recommended by NHS digital. Participants are asked to listen to one or two tracks daily for the initial 14 days, and as they find beneficial thereafter. They are then followed up, at 2 and 12 weeks, with their anxiety and depression scales (the GAD-7 and PHQ-9). The trial is a single site study that will take place at the Royal Free, with discharged patients in the community

ELIGIBILITY:
Inclusion criteria

* Over the age of 18
* Treated for Covid-19 at the Royal Free Hospital
* Capacity to consent AND
* At screening had a PHQ-2 score >=3 (positive) OR
* At screening had a TSQ score >= 6 (positive)

Exclusion criteria

* A current inpatient
* Participant on alternative trial that excludes being in a secondary trial
* Patient currently using alternative MBCT app tool
* Patients under 18 years old
* Background of psychotic illness
* Patient declined
* Patient unable to consent
* Underlying cognitive impairment which may impede ability to comply with the intervention
* Severe hearing impairment
* Current delirium
* Was an in-patient in intensive care during hospital stay
* Unable to contact patient via telephone on 2 attempts Patient is not registered with a GP. Unable to understand English proficiently enough to engage with the audio tracks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalised with Covid19 who have psychological symptoms 8 weeks after discharge. That is a >=6 on TSQ or >= 3 on PHQ9.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety as measured by generalised anxiety disorder score (GAD-7) scale | Day 14
  Generalised anxiety disorder score (GAD-7) scale. Score 0-21, with a higher score associated with greater anxiety symptoms. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. GAD-7 score at baseline will be controlled for.

SECONDARY OUTCOMES:
Depression as measured by the patient health questionnaire 9 (PHQ-9) | 14 days and week 12
  The Patient Health Questionnaire (PHQ-9) is a screening tool for the identification of depressive disorders, which has been validated for use in primary care. Each of the nine items in the questionnaire is based on the DSM diagnostic criteria for clinical depression. The PHQ-9 is scored out of 27 according to severity, where score of 5-9 indicates mild depression, 10-14 moderate, 15-19 moderately severe, and 20 or above severe depression.
Trauma as measured by Trauma screening questionnaire (TSQ) | 12 weeks
  The Trauma screening questionnaire (TSQ) is a 10 point scale used to identify symptoms of post traumatic stress disorder (PTSD), with a score between 0 and 10, with a score of 6 or higher scored as positive.
Anxiety as measured by generalised anxiety disorder score (GAD-7) scale | Week 12
  Generalised anxiety disorder score (GAD-7) scale. Score 0-21, with a higher score associated with greater anxiety symptoms. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. GAD-7 score at baseline will be controlled for.

OTHER OUTCOMES:
Risk associated with distress | Baseline analysis
  Risk factors for psychological distress from admission with Covid-19 will be collected, these will include, age, gender, ethnicity, length of hospital stay, oxygen requirement, co-morbidites, years of education, smoking status, occupation.
Qualitative analysis | Baseline
  Framework analysis. Qualitative feedback of patient experience. Semi structured interviews of a subset of patients will be performed to gain further insight into the patient experience. These will be analysed using a framework thematic analysis, to identify themes which will then be used to code the text.

CONTACTS AND LOCATIONS:
Overall Officials: Research and Development Manager, Study Chair — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: No